CLINICAL TRIAL: NCT04513444
Title: Phase II Study Aiming to Evaluate the Interest of Medical Hypnosis in Anxious Patients Treated by Radiotherapy
Brief Title: Interest of Medical Hypnosis in Anxious Patients Treated by Radiotherapy
Acronym: HYPNOMUSE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20 GENE 07
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumor
Keywords: Solid Tumor; Radiotherapy; Hypnosis; Anxiety; Music listening
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard arm (A): music listening therapy (Other)
  Interventions: Other: Relaxation with music listening during radiotherapy treatment:
- Experimental arm (B): music listening and hypnosis therapy (Experimental)
  Interventions: Other: Relaxation with music listening and medical hypnosis during radiotherapy treatment:

INTERVENTIONS:
Other: Relaxation with music listening and medical hypnosis during radiotherapy treatment: — * Music listening (According to the patient's wishes),
  * Hypnosis sessions with the hypnotherapist during the 1st, 2nd and 3rd radiotherapy session,
  * Self-hypnosis during the 4th and 5th radiotherapy session,
  * Questionnaires (STAI-Y and QLQ-C30) and numerical scales (anxiety and pain) will be completed by patients during radiotherapy consultations.
  Arms: Experimental arm (B): music listening and hypnosis therapy
Other: Relaxation with music listening during radiotherapy treatment: — * Music listening (According to the patient's wishes),
  * Questionnaires (STAI-Y and QLQ-C30) and numerical scales (anxiety and pain) will be completed by patients during radiotherapy consultations.
  Arms: Standard arm (A): music listening therapy

SUMMARY:
This phase II, randomized, non-comparative and monocentric study aims to evaluate the interest of medical hypnosis in the management of anxiety in patients who are moderately anxious, anxious or very anxious during their radiotherapy treatment.

45 patients will be randomized into the following arms:

* Arm A (standard): relaxation with music listening during radiotherapy treatment
* Arm B (experimental): relaxation with music listening and hypnosis during radiotherapy treatment

For the study each patient will be followed during 2 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of enrollment into the study.
2. Patient with localized or metastatic solid malignant tumor.
3. Patient being followed for the cancer pathology at IUCT-O and to receive, for the first time in the follow-up, treatment by radiotherapy (radiotherapy treatment should not have been initiated prior to inclusion in the study).
4. Patient for whom radiotherapy treatment includes at least 15 sessions of radiation therapy.
5. Patient defined as moderately anxious, anxious or very anxious after completing the STAI-Y self-assessment questionnaire (i.e. ≥ 46 score at inclusion).
6. ECOG patient ≤ 2.
7. Patient who signed informed consent prior to inclusion in the study and prior to any specific study procedures.
8. Patient affiliated to a Social Health Insurance in France.

Exclusion Criteria:

1. Patient doesn't understand the French language.
2. Patient with psychiatric disorders requiring antidepressant or antipsychotic treatment.
3. Patient with hearing problems.
4. Pregnant or breastfeeding women.
5. Any psychological, family, geographical or sociological condition that prevents compliance with the medical follow-up and/or procedures of the study protocol.
6. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-12-07 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with at least a 10-point decrease in anxiety score (evolution between the baseline and the 6th and last radiotherapy session) | 2 months for each patient
  Anxiety will be assessed using the STAI-Y questionnaire (Spielberger State-Trait Anxiety Inventory - State Anxiety form).

SECONDARY OUTCOMES:
Anxiety assessed using a numerical scale from 0 to 10 (0 being "not at all anxious" and 10 being "extremely anxious") | 2 months for each patient
Quality of life assessed using the EORTC (European Organization for Research and Treatment of Cancer) Quality of life questionnaire (QLQ-C30). | 2 months for each patient
  Changes in quality of life from baseline will be assessed in the classroom according to the recommendations of the literature (Osoba, JCO).

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse, France